CLINICAL TRIAL: NCT06125132
Title: Evaluation of 2-year Clinical Performance of Two Different Single Color Universal Composite Resin Restorative Materials: A Double-blind Prospective Randomized Controlled Trial.
Brief Title: Evaluation of 2-year Clinical Performance of Two Different Single Color Universal Composite Resin Restorative Materials.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Leyla Kerimova, lecturer, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-KA22/25
Record Dates: First submitted 2023-10-27; First posted 2023-11-09 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Tooth Discoloration; Tooth Wear
Keywords: one-shade composites; single-shade composites; universal composites
MeSH Terms: conditions — Tooth Discoloration; Tooth Wear

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- OMNICHROMA one shade composite (Active Comparator): a one-shade composite resin as experimental group
  Interventions: Procedure: Restoration with-tooth colored material
- Zen Chroma one shade composite (Active Comparator): a one-shade composite resin as experimental group
  Interventions: Procedure: Restoration with-tooth colored material
- Filtek Z250 multi shade composite (Active Comparator): a multi-shade composite resin as control group
  Interventions: Procedure: Restoration with-tooth colored material

INTERVENTIONS:
Procedure: Restoration with-tooth colored material — Restoration of abrasions with different composite resin materials

SUMMARY:
Dentists have recently preferred to use composite materials and restorative techniques that allow the use of simplified clinical protocols in order to reduce the time the patient spends in the dentist's chair and minimize technical sensitivity. Color selection in the clinic is a very sensitive process and is affected by environmental factors and operator-related variables. This has led to the development of single-color universal composite resins that aim to facilitate color selection. These materials have a universal opacity and several Vita shades and are recommended by manufacturers to be used in a single color layer that can match different tooth colors. In recent years, monochromatic universal composites have been developed that are supposed to be compatible with all Vita Classic Scale shades from A1 to D4. Manufacturers report that single-color universal composites can be applied to teeth of all colors without using the layering technique using different color composites.

Therefore, the aim of this study is to compare the clinical performance of 2 different single-color universal composite resin materials (OMNICHROMA and Zenchroma) in the restoration of non-carious cervical lesions with the control group (Filtek Z250, 3M), which is a multi-color composite resin material, using modified US Public Health Service (USPHS) and World Dental Federation (FDI) criteria.

DETAILED DESCRIPTION:
Dentists have recently preferred to use composite materials and restorative techniques that allow the use of simplified clinical protocols in order to reduce the time the patient spends in the dentist's chair and minimize technical sensitivity. Color selection in the clinic is a very sensitive process and is affected by environmental factors and operator-related variables. This has led to the development of single-color universal composite resins that aim to facilitate color selection. These materials have a universal opacity and several Vita shades and are recommended by manufacturers to be used in a single color layer that can match different tooth colors. In recent years, monochromatic universal composites have been developed that are supposed to be compatible with all Vita Classic Scale shades from A1 to D4. Manufacturers report that single-color universal composites can be applied to teeth of all colors without using the layering technique using different color composites.

OMNICHROMA (Tokuyama Dental) is the first universal composite resin restorative material that is claimed to aesthetically match every tooth color from A1 to D4 in a single shade. The manufacturer declares that OMNICHROMA, with its equally sized supra-nano spherical filler (260 nm spherical silicon dioxide-Zzirconium dioxide), adapts to each of the 16 VITA classic colors thanks to Smart Chromatic Technology.

Zenchroma (President Dental) is a hybrid composite material containing an ultra-thin, radiopaque glass filler. The manufacturer declares that the filling color perfectly adapts to the tooth structure with its chameleon effect.

As we know, there is no study investigating the clinical performance of these two universal composites. The aim of this study is to compare the clinical performance of 2 different single-color universal composite resin materials (OMNICHROMA and Zenchroma) in the restoration of non-carious cervical lesions with the control group (Filtek Z250, 3M), which is a multi-color composite resin material, using modified USPHS and FDI criteria.

In this study, two different null hypotheses were established. The first null hypothesis of this study is; It is concluded that there is no difference between 2 different single color universal composite resin materials (OMNICHROMA and Zenchroma) in terms of clinical performance in restorations of non-carious cervical lesions. The second null hypothesis of the study is that universal composite resin materials are not different from the control group, multicolored composite resin (Filtek Z250, 3M), in terms of clinical performance in restorations of non-carious cervical lesions.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 teeth with cervical abrasion
* Volunteerily enrolling

Exclusion Criteria:

* No bruxism
* No carious formation in worn teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical performance according to the modified United States Public Health Service criteria | 6,12,18, 24 and 36 months
  Retention, marginal discoloration, marginal adaptation, secondary caries and postoperative sensitivity will be scored as Alpha (the best), Bravo (acceptable) and Charlie (unacceptable).

SECONDARY OUTCOMES:
Clinical performance of restorations according to the World Dental Organization criteria | 6,12,18, 24 and 36 months
  Retention, marginal discoloration, marginal adaptation, secondary caries and postoperative sensitivity will be scored as 1) clinically excellent, 2) clinicallay good, 3) clinically sufficient, 4) clinically unsatisfactory and 5) clinically poor

CONTACTS AND LOCATIONS:
Overall Officials: Kıvanç Yamanel, PHD, Study Director — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] de Abreu JLB, Sampaio CS, Benalcazar Jalkh EB, Hirata R. Analysis of the color matching of universal resin composites in anterior restorations. J Esthet Restor Dent. 2021 Mar;33(2):269-276. doi: 10.1111/jerd.12659. Epub 2020 Sep 29. PMID 32989879
- [Background] Durand LB, Ruiz-Lopez J, Perez BG, Ionescu AM, Carrillo-Perez F, Ghinea R, Perez MM. Color, lightness, chroma, hue, and translucency adjustment potential of resin composites using CIEDE2000 color difference formula. J Esthet Restor Dent. 2021 Sep;33(6):836-843. doi: 10.1111/jerd.12689. Epub 2020 Dec 7. PMID 33283966
- [Background] Iyer RS, Babani VR, Yaman P, Dennison J. Color match using instrumental and visual methods for single, group, and multi-shade composite resins. J Esthet Restor Dent. 2021 Mar;33(2):394-400. doi: 10.1111/jerd.12621. Epub 2020 Aug 25. PMID 32844567
- [Background] Kobayashi S, Nakajima M, Furusawa K, Tichy A, Hosaka K, Tagami J. Color adjustment potential of single-shade resin composite to various-shade human teeth: Effect of structural color phenomenon. Dent Mater J. 2021 Jul 31;40(4):1033-1040. doi: 10.4012/dmj.2020-364. Epub 2021 Apr 20. PMID 33883353
- See also: Zen Chroma Universal Composite — http://www.presidentdental.com